CLINICAL TRIAL: NCT05066217
Title: Multicenter, Randomized, Double-blind, Placebo-controlled Trial of Clemizole HCl as Adjunctive Therapy in Patients With Lennox-Gastaut Syndrome
Brief Title: An Efficacy and Safety Study of Clemizole HCl in Patients With Lennox-Gastaut Syndrome
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Epygenix (Industry)
Collaborators: Harmony Biosciences Management, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EPX-100-003
Record Dates: First submitted 2021-09-23; First posted 2021-10-04 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Lennox Gastaut Syndrome
Keywords: Lennox Gastaut Syndrome; Lennox-Gastaut Syndrome; LGS; Clemizole HCl; Seizure
MeSH Terms: conditions — Lennox Gastaut Syndrome; Seizures

STUDY DESIGN:
Intervention Model Description: Patients are randomized 1:1 to clemizole HCl (EPX-100) or placebo.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Participants will receive their first dose of study drug following randomization.
  Interventions: Drug: Placebo
- Double-blind clemizole HCl (Experimental): Participants will receive their first dose of study drug following randomization.
  Interventions: Drug: Clemizole HCl
- Open-label clemizole HCl (Experimental): Eligible participants who complete the DB Period will have the option to continue in the OLE Period, during which they will receive clemizole HCl for up to 3 years.
  Interventions: Drug: Clemizole HCl; Drug: Placebo

INTERVENTIONS:
Drug: Clemizole HCl — Clemizole HCl will be administered as an oral solution.
  Other Names: EPX-100
  Arms: Double-blind clemizole HCl; Open-label clemizole HCl
Drug: Placebo — Placebo will be administered as an oral solution.
  Arms: Open-label clemizole HCl; Placebo

SUMMARY:
This is a multicenter, Phase 3, randomized, double-blind, placebo-controlled study designed to evaluate the efficacy and safety of clemizole HCL (EPX-100) as adjunctive therapy in children and adult participants with Lennox-Gastaut syndrome (LGS).

DETAILED DESCRIPTION:
This is a multicenter, Phase 3, randomized, double-blind, placebo-controlled study designed to evaluate the efficacy and safety of clemizole HCl as adjunctive therapy in children and adult participants with LGS.

The study will consist of an Observational Period, a Double-Blind (DB) Period, and an optional Open-Label Extension (OLE) Period.

ELIGIBILITY:
Key Inclusion Criteria:

1. Males or females, ages ≥2 to ≤55 years, at the time of Screening.
2. Participant/parent/legal authorized representative (LAR) willing and able to give written informed consent/assent.
3. Diagnosis of LGS, including:

   * Evidence of at least one type of countable major motor seizure.
   * History of electroencephalogram (EEG) consistent with LGS (abnormal background activity, and one of the following: 1) slow spike-wave discharges [<2.5 Hz], or 2) paroxysmal fast activity during sleep).
   * Abnormal cognitive development.
   * Onset of seizures at 11 years of age or younger.

Key Exclusion Criteria:

1. Known sensitivity, allergy, or previous exposure to clemizole HCl.
2. Known history of long QT syndrome or any significant history of a serious abnormality of the electrocardiogram (ECG) (e.g., recent myocardial infarction, clinically significant arrhythmia).
3. Family history of sudden cardiac death, unexplained death, or death from a primary dysrhythmia potentially associated with QT prolongation in any family member.
4. Seizures secondary to illicit drug or alcohol use, infection, neoplasm, demyelinating disease, degenerative neurological disease, or progressive central nervous system disease, metabolic illness, recent anoxic episode within the last 6 months requiring resuscitation, or progressive degenerative disease or any other condition, which in the opinion of the investigator, could affect seizure control.
5. Epilepsy surgery planned during the study or epilepsy surgery within 6 months prior to Screening.
6. Concomitant use of fenfluramine.
7. Prior or concomitant use of lorcaserin.

Ages: 2 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 260 (Estimated)
Dates: Start 2025-04-09 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2029-11-01 (Estimated)

PRIMARY OUTCOMES:
Percent Change in CMMS-28 | From Baseline Period up to 16 weeks
  Percent change in CMMS-28 from the Baseline Period through the end of the DB Period

SECONDARY OUTCOMES:
Proportion of Participants with ≥50% Reduction in CMMS-28 | From Baseline Period up to 16 weeks
  Proportion of participants with ≥50% reduction in CMMS-28 from the Baseline Period through the end of the DB Period
Percent Change in CMMS-28 Seizure-free Days | From Baseline Period up to 16 weeks
  Percent change in CMMS-28 seizure-free days from the Baseline Period through the end of the DB Period
Clinical Global Impression of Change (CGI-C) Score | Week 16
  CGI-C score at the end of the DB Period
Caregiver Global Impression of Change (CaGI-C) Score | Week 16
  CaGI-C score at the end of the DB Period
Caregiver Global Impression of Change in Seizure Intensity/Duration (CaGI-CSID) Score | Week 16
  CaGI-CSID score at the end of the DB Period
Change in Quality of Life Inventory (QI)-Disability Score | From Baseline Period up to 16 weeks
  Change in QI-disability score from Baseline to the end of the DB Period
Percent Change per 28 Days in the Number of Seizure Free Days | From Baseline Period up to 16 weeks
  Percent change per 28 days in the number of seizure-free days (based on all seizure types) from the Baseline Period through the end of the DB Period
Percent Change in CMMS-28 | From Baseline Period up to 12 weeks
  Percent change in CMMS-28 from the Baseline Period through the end of the DB Maintenance Phase only
Proportion of Participants with ≥50% Reduction in CMMS-28 | From Baseline Period up to 12 weeks
  Proportion of participants with ≥50% reduction in CMMS-28 from the Baseline Period through the end of the DB Maintenance Phase only
Incidence of Treatment-Emergent Adverse Events (TEAEs) | From the first dose administration of study drug up to end of the study, approximately up to 172 weeks
  Incidence of TEAEs will be compared among the treatment groups

CONTACTS AND LOCATIONS:
Overall Officials: Amit Ray, MD, Study Director — Harmony Biosciences Management, Inc.
Locations (4):
- United States (4):
  - Rare Disease Research, Kissimmee, Florida
  - Minnesota Epilepsy Group, P.A., Roseville, Minnesota
  - Neurology Center for Epilepsy and Seizures, Marlboro, New Jersey
  - On-Site Clinical Solution, Charlotte, North Carolina

IPD SHARING:
Plan to Share IPD: No